CLINICAL TRIAL: NCT03547973
Title: A Phase II Open-Label Study of Sacituzumab Govitecan in Unresectable Locally Advanced/Metastatic Urothelial Cancer
Brief Title: Study of Sacituzumab Govitecan in Participants With Urothelial Cancer That Cannot Be Removed or Has Spread
Acronym: TROPHY U-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMMU-132-06; 2023-508302-24 (Other: European Medicines Agency)
Record Dates: First submitted 2018-04-26; First posted 2018-06-06 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Urothelial Cancer
MeSH Terms: interventions — sacituzumab govitecan; pembrolizumab; Cisplatin; avelumab; zimberelimab; Carboplatin; Gemcitabine; enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Cohort 1: Sacituzumab Govitecan-hziy (SG) (Experimental): Participants with urothelial cancer (UC) previously treated with platinum-based and/or checkpoint inhibitors (CPIs) will receive SG 10 mg/kg intravenously (IV) on Days 1 and 8 of a 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Cohort 2: SG (Experimental): Participants with UC who are ineligible for platinum-based therapy and failed therapy with previous immune CPI therapy will receive SG 10 mg/kg intravenously on Days 1 and 8 of a 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Cohort 3: SG + Pembrolizumab (Experimental): Participants who have had progression or recurrence of UC following a platinum-containing regimen in the metastatic setting, or progression or recurrence of UC within 12 months of completion of platinum-based therapy as neoadjuvant or adjuvant therapy will receive SG 10 mg/kg intravenously on Days 1 and 8 of a 21-day cycle and pembrolizumab at the standard approved dose (200 mg) only on Day 1 of a 21-day cycle. Lower doses of SG may be tested based on dose-limiting toxicities (DLTs) observed to determine the Recommended Phase 2 Dose (RP2D) of SG in combination with pembrolizumab.
  Interventions: Drug: Sacituzumab Govitecan-hziy; Drug: Pembrolizumab
- Cohort 4: SG + Cisplatin + Avelumab (Dose Escalation Phase) (Experimental): Participants with UC who have never received therapy with platinum in the metastatic setting or for unresectable locally advanced disease will first receive cisplatin (either at 70 mg/m^2 on Day 1 of a 21-day cycle or at a split dose of 35 mg/m^2 on Days 1 and 8 of a 21-day cycle with a maximum body surface area of 2) and sacituzumab govitecan-hziy with maximum dose of 10 mg/kg intravenously on Days 1 and 8 of a 21-day cycle for up to 6 cycles. Based on DLTs observed, two additional lower doses may be tested to determine RP2D of sacituzumab govitecan-hziy in combination with cisplatin. If premature termination of 1 agent occurs due to toxicity, the other agent may be continued to complete up to 6 cycles of therapy. For participants who have not progressed, maintenance therapy will begin with infusions of avelumab 800 mg every 2 weeks beginning on Cycle 1, Day 1 and every 2 weeks thereafter and sacituzumab govitecan-hziy 10 mg/kg on Days 1 and 8 every 21 days.
  Interventions: Drug: Sacituzumab Govitecan-hziy; Drug: Cisplatin; Drug: Avelumab
- Cohort 4: SG + Cisplatin + Zimberelimab (ZIM) (Dose Expansion Phase) (Experimental): Participants with UC who have never received therapy with platinum in the metastatic setting or for unresectable locally advanced disease will first receive cisplatin (either at 70 mg/m^2 on Day 1 of a 21-day cycle or at a split dose of 35 mg/m^2 on Days 1 and 8 of a 21-day cycle with a maximum body surface area of 2) and sacituzumab govitecan-hziy with maximum dose of 10 mg/kg intravenously on Days 1 and 8 of a 21-day cycle for up to 6 cycles. If premature termination of 1 agent occurs due to toxicity, the other agent may be continued to complete up to 6 cycles of therapy. For participants who have not progressed, maintenance therapy will begin with infusions of sacituzumab govitecan-hziy 10 mg/kg on Days 1 and 8 every 21 days and zimberelimab 360 mg every 3 weeks (Day 1 of a 21-day cycle).
  Interventions: Drug: Sacituzumab Govitecan-hziy; Drug: Cisplatin; Drug: Zimberelimab
- Cohort 5 (Arm 1): SG + ZIM (Experimental): Participants in Cohort 5 will have completed 4 to 6 cycles of gemcitabine (GEM) + cisplatin therapy without PD prior to study entry. The safety lead-in will be conducted, in 6 to 8 participants (treated with SG 10 mg/kg IV on Day 1 and Day 8 of a 21-day cycle + ZIM 360 mg IV every 3 weeks on a 21-day cycle). Upon completion of the safety lead-in, participants will receive SG 10 mg/kg IV on Days 1 and 8 of a 21-day cycle followed by ZIM 360 mg IV, every 3 weeks (Q3W) (Day 1 of a 21-day cycle) until PD, unacceptable toxicity, or loss of clinical benefit. participants who must discontinue 1 agent may continue the other until PD, unacceptable toxicity, or loss of clinical benefit.
  Interventions: Drug: Sacituzumab Govitecan-hziy; Drug: Zimberelimab
- Cohort 5 (Arm 2): Avelumab (Experimental): Participants in Cohort 5 will have completed 4 to 6 cycles of gemcitabine (GEM) + cisplatin therapy without PD prior to study entry. The safety lead-in will be conducted, in 6 to 8 participants (treated with SG 10 mg/kg IV on Day 1 and Day 8 of a 21-day cycle + ZIM 360 mg IV every 3 weeks on a 21-day cycle). Upon completion of the safety lead-in, participants will be randomized to receive avelumab 800 mg IV every 2 weeks (Q2W) until PD, unacceptable toxicity, or loss of clinical benefit.
  Interventions: Drug: Avelumab
- Cohort 5 (Arm 3): ZIM (Experimental): Participants in Cohort 5 will have completed 4 to 6 cycles of gemcitabine (GEM) + cisplatin therapy without PD prior to study entry. The safety lead-in will be conducted, in 6 to 8 participants (treated with SG 10 mg/kg IV on Day 1 and Day 8 of a 21-day cycle + ZIM 360 mg IV every 3 weeks on a 21-day cycle).
  Upon completion of the safety lead-in, participants will be randomized to receive ZIM 360 mg IV Q3W (Day
  1 of a 21-day cycle) until PD, unacceptable toxicity, or loss of clinical benefit.
  Interventions: Drug: Zimberelimab
- Cohort 6 (Arm 1): SG (Experimental): Upon completion of the safety lead-in, participants in Cohort 6 will be randomized and SG will be administered in cisplatin-ineligible participants who have never received therapy in the metastatic setting or for unresectable locally advanced disease. Treatment may be discontinued at any time, but participants will continue to be followed for tumor response until progression is documented, and alternate therapy is initiated. If participants discontinue therapy before evidence of radiologic progression, imaging should continue until radiologic progression is documented, if feasible.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Cohort 6 (Arm 2): SG + ZIM (Experimental): Upon completion of the safety lead-in, participants in Cohort 6 will be randomized and SG in combination with ZIM will be administered in cisplatin-ineligible participants who have never received therapy in the metastatic setting or for unresectable locally advanced disease. The standard approved dose of SG will be used in combination with ZIM. Treatment may be discontinued at any time, but participants will continue to be followed for tumor response until progression is documented or alternate therapy is initiated. If participants discontinue therapy before evidence of radiologic progression, imaging should continue until radiologic progression is documented, if feasible.
  Interventions: Drug: Sacituzumab Govitecan-hziy; Drug: Zimberelimab
- Cohort 6 (Arm 3): SG + ZIM + Domvanalimab (DOM) (Experimental): Upon completion of the safety lead-in, participants in Cohort 6 will be randomized and SG in combination with ZIM and DOM will be administered in cisplatin-ineligible participants who have never received therapy in the metastatic setting or for unresectable locally advanced disease.
  Interventions: Drug: Sacituzumab Govitecan-hziy; Drug: Zimberelimab; Drug: Domvanalimab
- Cohort 6 (Arm 4): Carboplatin (CARBO) + Gemcitabine (GEM) (Experimental): Upon completion of the safety lead-in, participants in Cohort 6 will be randomized and CARBO in combination with GEM will be administered in cisplatin-ineligible participants who have never received therapy in the metastatic setting or for unresectable locally advanced disease. Participants without disease progression as assessed by the investigator after completion of 4 to 6 cycles of therapy may continue with maintenance therapy (avelumab 800 mg every 2 weeks) until loss of clinical benefit.
  Interventions: Drug: Avelumab; Drug: Carboplatin; Drug: Gemcitabine
- Cohort 7 (Phase 1: Safety Lad-in and Dose Expansion): SG + Enfortumab Vedotin (EV) + ZIM (Experimental): In the safety lead-in phase, participants will receive a starting dose level of SG 7.5 mg/kg IV and starting dose level of EV 1.25 mg/kg IV will be administered on Days 1 and 8 of each 21-day cycle and ZIM 360 mg IV will be administered on Day 1 of each 21-day cycle.
  In dose-expansion, participants will receive SG IV and EV IV at the RP2Ds on Days 1 and 8 of each 21-day cycle and ZIM 360 mg IV on Day 1 of each 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy; Drug: Zimberelimab; Drug: Enfortumab Vedotin
- Cohort 7 (Phase 2: Arm 1): SG + EV + ZIM (Experimental): Upon completion of the Cohort 7 dose-expansion phase, participants will receive SG IV at the RP2D in combination with EV IV at the RP2D, and ZIM 360 mg IV until PD, unacceptable toxicity, or loss of clinical benefit.
  Interventions: Drug: Sacituzumab Govitecan-hziy; Drug: Zimberelimab; Drug: Enfortumab Vedotin
- Cohort 7 (Phase 2: Arm 2): EV + ZIM (Experimental): Upon completion of the Cohort 7 dose-expansion phase, participants will receive EV 1.25 mg/kg IV and ZIM 360 mg IV.
  Interventions: Drug: Zimberelimab; Drug: Enfortumab Vedotin
- Cohort 7 (Phase 2: Arm 3): Optional Dose Optimization SG + EV + ZIM (Experimental): Upon completion of the Cohort 7 dose-expansion phase, participants will receive SG IV at 1 dose level below the RP2D in combination with EV 1.25 mg/kg IV and ZIM 360 mg IV.
  Interventions: Drug: Sacituzumab Govitecan-hziy; Drug: Zimberelimab; Drug: Enfortumab Vedotin

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy — Administered intravenously.
  Other Names: IMMU-132; Trodelvy™
  Arms: Cohort 1: Sacituzumab Govitecan-hziy (SG); Cohort 2: SG; Cohort 3: SG + Pembrolizumab; Cohort 4: SG + Cisplatin + Avelumab (Dose Escalation Phase); Cohort 4: SG + Cisplatin + Zimberelimab (ZIM) (Dose Expansion Phase); Cohort 5 (Arm 1): SG + ZIM; Cohort 6 (Arm 1): SG; Cohort 6 (Arm 2): SG + ZIM; Cohort 6 (Arm 3): SG + ZIM + Domvanalimab (DOM); Cohort 7 (Phase 1: Safety Lad-in and Dose Expansion): SG + Enfortumab Vedotin (EV) + ZIM; Cohort 7 (Phase 2: Arm 1): SG + EV + ZIM; Cohort 7 (Phase 2: Arm 3): Optional Dose Optimization SG + EV + ZIM
Drug: Pembrolizumab — Administered per package insert
  Other Names: KEYTRUDA®
  Arms: Cohort 3: SG + Pembrolizumab
Drug: Cisplatin — Administered per package insert
  Arms: Cohort 4: SG + Cisplatin + Avelumab (Dose Escalation Phase); Cohort 4: SG + Cisplatin + Zimberelimab (ZIM) (Dose Expansion Phase)
Drug: Avelumab — Administered per package insert
  Other Names: BAVENCIO®
  Arms: Cohort 4: SG + Cisplatin + Avelumab (Dose Escalation Phase); Cohort 5 (Arm 2): Avelumab; Cohort 6 (Arm 4): Carboplatin (CARBO) + Gemcitabine (GEM)
Drug: Zimberelimab — Administered intravenously
  Arms: Cohort 4: SG + Cisplatin + Zimberelimab (ZIM) (Dose Expansion Phase); Cohort 5 (Arm 1): SG + ZIM; Cohort 5 (Arm 3): ZIM; Cohort 6 (Arm 2): SG + ZIM; Cohort 6 (Arm 3): SG + ZIM + Domvanalimab (DOM); Cohort 7 (Phase 1: Safety Lad-in and Dose Expansion): SG + Enfortumab Vedotin (EV) + ZIM; Cohort 7 (Phase 2: Arm 1): SG + EV + ZIM; Cohort 7 (Phase 2: Arm 2): EV + ZIM; Cohort 7 (Phase 2: Arm 3): Optional Dose Optimization SG + EV + ZIM
Drug: Carboplatin — Administered per package insert
  Arms: Cohort 6 (Arm 4): Carboplatin (CARBO) + Gemcitabine (GEM)
Drug: Gemcitabine — Administered per package insert
  Arms: Cohort 6 (Arm 4): Carboplatin (CARBO) + Gemcitabine (GEM)
Drug: Domvanalimab — Administered intravenously
  Arms: Cohort 6 (Arm 3): SG + ZIM + Domvanalimab (DOM)
Drug: Enfortumab Vedotin — Administered intravenously
  Arms: Cohort 7 (Phase 1: Safety Lad-in and Dose Expansion): SG + Enfortumab Vedotin (EV) + ZIM; Cohort 7 (Phase 2: Arm 1): SG + EV + ZIM; Cohort 7 (Phase 2: Arm 2): EV + ZIM; Cohort 7 (Phase 2: Arm 3): Optional Dose Optimization SG + EV + ZIM

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of sacituzumab govitecan-hziy monotherapy and with novel combinations in participants with metastatic urothelial cancer (mUC).

DETAILED DESCRIPTION:
Non-Randomized for Cohorts 1,2,3, and 4; Randomized for Cohorts 5, 6, and 7. Cohort 5 has been cancelled, effective December 2023.

ELIGIBILITY:
Key Inclusion Criteria:

Inclusion Criteria for All Cohorts:

* Female or male individuals, ≥ 18 years of age (19 Years old for South Korea).
* Eastern Cooperative Oncology Group (ECOG) Performance status score of 0 or 1.
* Adequate renal and hepatic function.
* Adequate hematologic parameters without transfusional support.
* Individuals must have a 3-month life expectancy.

Additional Inclusion Criteria for Cohorts 1 to 6:

* Cohort 1: Have had progression or recurrence of urothelial cancer following receipt of platinum-containing regimen (cisplatin or carboplatin):

  1. Received a first-line platinum-containing regimen in the metastatic setting or for inoperable locally advanced disease;
  2. Or received neo/adjuvant platinum-containing therapy for localized muscle-invasive urothelial cancer, with recurrence/progression ≤12 months following completion of therapy.
* Cohort 1: In addition to above criterion, have had progression or recurrence of urothelial cancer following receipt of an Anti-programmed Cell Death Protein 1 (anti-PD-1)/ Anti-programmed Death Ligand 1 (PD-L1) therapy.
* Cohort 2: Were ineligible for platinum-based therapy for first line metastatic disease and have had progression or recurrence of urothelial cancer after a first-line therapy for metastatic disease with anti-PD-1/PD-L1 therapy. Individual may not have received any platinum for treatment of recurrent, metastatic or advanced disease.
* Cohort 3: Progression or recurrence of UC following a platinum containing regimen in the metastatic setting, or progression or recurrence of UC within 12 months of completion of platinum-based therapy as neoadjuvant or adjuvant therapy.
* Cohort 4: Individual has not received any platinum-based chemotherapy in the metastatic or unresectable locally advanced setting. Creatinine clearance of at least 50 mL/min calculated by Cockcroft-Gault formula or another validated tool. For individuals receiving cisplatin at 70 mg/m^2 on Day 1 of every 21-day cycle, a creatinine clearance of least 60 mL/min calculated by Cockcroft -Gault formula or another validated tool is required. Individuals with creatinine clearance between 50 to 59 mL/min are to receive a split dose of cisplatin (35 mg/m^2 Day 1 and Day 8 of every 21-day cycle).
* Cohorts 4, 5, 6: Archival tumor tissue comprising muscle-invasive or metastatic urothelial carcinoma, or a biopsy of metastatic urothelial carcinoma.
* Cohort 5: Individuals received at least 4 cycles and no more than 6 cycles of GEM + cisplatin. No other chemotherapy regimens are allowed in this cohort, with the exception of prior adjuvant or neoadjuvant systemic therapy with curative intent after > 12 months from completion of therapy.
* No evidence of progressive disease following completion of first-line chemotherapy (ie, CR, PR, or SD per RECIST v1.1 guidelines as per investigator).
* Treatment-free interval of 4 to 10 weeks since the last dose of chemotherapy.
* Cohort 6: Cis-ineligible and no prior therapy for metastatic disease or for unresectable locally advanced disease. Checkpoint inhibitor therapy naïve or >12 months from completion of adjuvant therapy are permitted.
* Cohorts 4 and 6: Have measurable disease by CT or MRI as per RECIST 1.1 criteria. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Cohorts 1, 2, 3 and 5: Creatinine clearance ≥ 30 mL/min as calculated by the Cockcroft-Gault formula unless otherwise specified

Additional Inclusion Criteria for Cohort 7:

* No prior systemic therapy for locally advanced or metastatic UC. Therapy in the curative setting is allowed provided recurrence is > 12 months since the last dose of systemic therapy.
* Archival tumor tissue comprising muscle-invasive or metastatic urothelial carcinoma, or a biopsy of metastatic urothelial carcinoma.
* Have measurable disease by CT or MRI as per RECIST 1.1 criteria. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

Key Exclusion Criteria:

Exclusion Criteria for All cohorts:

* Females who are pregnant or lactating.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has an active second malignancy.
* Has known active Hepatitis B or Hepatitis C.
* Has other concurrent medical or psychiatric conditions.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has an active second malignancy.

Additional Exclusion Criteria for Cohorts 1 to 6:

* For Cohort 5: Alopecia, sensory neuropathy Grade ≤2 is acceptable, or other Grade << 2 adverse events not constituting a safety risk based on the investigator's judgment are acceptable.
* Cohort 3: Has received anti-PD-1/PD-L1 therapy previously.
* Cohorts 3 to 6: Has an active autoimmune disease that required systemic treatment in past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Cohorts 3 to 6: Has received a live vaccine within 30 days prior to the first dose of study drug(s), has history or evidence of interstitial lung disease (ILD) or non-infectious pneumonitis.
* Cohort 4: Refractory to platinum (i.e., relapsed ≤ 12 months after completion of chemotherapy) in the neoadjuvant/adjuvant setting.
* Cohorts 4, 5, and 6: For individuals who received prior CPI, a treatment-free interval >12 months between the last treatment administration and the date of recurrence is required.

Additional Exclusion Criteria for Cohort 7:

* Have had a prior anticancer therapy within 12 months prior to C1D1 or prior radiation therapy within 2 weeks prior to C1D1. Individuals participating in observational studies are eligible. Use of other investigational drugs (drugs not marketed for any indication) within 28 days or 5 half-lives (whichever is longer) of first dose of investigational product.
* Have a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Have a Child-Pugh score of B or C.
* Individuals with uncontrolled diabetes.
* Have active keratitis or corneal ulcerations.
* Participants with ongoing sensory or motor neuropathy Grade ≥ 2.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 827 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) Based on Central Review by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Criteria (Cohorts 1 to 4 and 6) | Up to Survival Follow-up Visit (maximum of 2 years after Safety Follow-up Visit (30 days after last dose date))
  ORR will be defined as the rate of the best overall response as Complete Response (CR) or Partial Response (PR) and based on central review by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) criteria.
Progression free survival (PFS) Based on Central Review by RECIST 1.1 criteria (Cohort 5) | Up to Survival Follow-up Visit (maximum of 2 years after Safety Follow-up Visit (30 days after last dose date))
  PFS will be defined as the time from first dose until objective tumor progression, as assessed based on central review, or death, whichever comes first.
ORR Based on Investigator Review by RECIST 1.1 Criteria (Cohort 7) | Up to Survival Follow-up Visit (maximum of 2 years after Safety Follow-up Visit (30 days after last dose date))
  ORR will be defined as the rate of the best overall response as Complete Response (CR) or Partial Response (PR) and based on investigator review by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) criteria.
Percentage of Participants Experiencing Treatment Emergent Adverse Events (TEAEs) (Cohort 7) | First dose date up to last dose date plus 30 days (approximately 3 years)
Percentage of Participants Experiencing any Clinically Significant Laboratory Abnormalities (Cohort 7) | First dose date up to last dose date plus 30 days (approximately 3 years)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to Survival Follow-up Visit (maximum of 2 years after Safety Follow-up Visit (30 days after last dose date))
  ORR will be defined as the rate of the best overall response as CR or PR and based on investigator review by RECIST 1.1 criteria for cohorts 3, 4, 6, and 7. ORR will also be evaluated based on investigator review by Modified RECIST 1.1 for Immune-Based Therapeutics (iRECIST 1.1) for Cohorts 3, 4, 6, and 7.
Duration of Response (DOR) | Up to Survival Follow-up Visit (maximum of 2 years after Safety Follow-up Visit (30 days after last dose date))
  DOR will be calculated from the date of the first evaluation showing documented response, PR, or CR, to the date of the first disease progression or death and based on central and investigator review by RECIST 1.1 criteria for all cohorts. DOR will also be evaluated based on investigator review by iRECIST 1.1 for Cohorts 3, 4, 6, and 7.
Progression-Free Survival (PFS) | Up to Survival Follow-up Visit (maximum of 2 years after Safety Follow-up Visit (30 days after last dose date))
  PFS is defined as the time from the first dose (Cohorts 1 through 4) or randomization date (Cohorts 5 through 7) until objective tumor progression,or death, whichever comes first and based on central and investigator review by RECIST 1.1 criteria for all cohorts. PFS will also be evaluated based on investigator review by iRECIST 1.1 for Cohorts 3, 4, 6, and 7.
Overall Survival (OS) | Up to Survival Follow-up Visit (maximum of 2 years after Safety Follow-up Visit (30 days after last dose date))
  OS will be measured from the date of first dose (Cohorts 1 through 4) or randomization date (Cohorts 5 through 7) to death from any cause.
Clinical Benefit Rate (CBR) | Up to Survival Follow-up Visit (maximum of 2 years after Safety Follow-up Visit (30 days after last dose date))
  CBR is defined as CR + PR + Stable Disease (SD) for at least 6 months and based on central and investigator review by RECIST 1.1 criteria for Cohorts 3, 4, 6, and 7. CBR will also be evaluated based on investigator review by iRECIST 1.1 for Cohorts 3, 4, 6, and 7.
Percentage of Participants Experiencing Treatment Emergent Adverse Events (TEAEs) (Cohorts 3, 4, 5, and 6) | First dose date up to last dose date plus 30 days (approximately 3 years)
Percentage of Participants Experiencing any Clinically Significant Laboratory Abnormalities (Cohorts 3, 4, 5, and 6) | First dose date up to last dose date plus 30 days (approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (135):
- United States (37):
  - The University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Woodlands Medical Specialists, PA, Pensacola, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Southern Illinois University School of Medicine, Simmons Cancer Institute, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Norton Cancer Institute, Downtown, Louisville, Kentucky
  - Maryland Oncology Hematology, P.A., Brandywine, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Oncology Hematology West PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Precision Cancer Research / New Mexico Oncology & Hematology Consultants, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Drug Shipping Address: New York-Presbyterian Hospital, New York, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - St. Luke's Hosptial - Bethlehem Campus, Easton, Pennsylvania
  - Medical University of Southern Carolina, Charleston, South Carolina
  - Thompson Oncology Group - Knoxville West, Knoxville, Tennessee
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Houston Methodist Hospital, Houston Methodist Cancer Center, Houston, Texas
  - Mays Cancer Center, San Antonio, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - University of Utah - Huntsman Cancer Hospital (IP Shipping Address), Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Oncology Associates, Hampton, Virginia
  - Oncology Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Roanoke, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
- France (21):
  - Centre Hospitalier Regional Universitaire (CHRU) de Besancon, Hopital Jean Minjoz, Besançon
  - Hopital Saint Andre (CHU de Bordeaux), Bordeaux
  - Centre Hospitalier Regional Universitaire Brest, Brest
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Departmental (CHD) Vendee, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Universitaire De Nimes - Hopital Universitaire Caremeau, Nîmes
  - Hopital European Georges-Pompidou (HEGP), Paris
  - Groupement Hospitalier Pitie-Salpetriere, Paris
  - Hopital Cochin, Paris
  - Centre Hospitalier Prive Saint-Gregoire, Rennes
  - Centre Eugene Marquis, Rennes
  - CHU de Rouen, Rouen
  - Hospitaux Universitaires de Strasbourg - Hopital Civil, Strasbourg
  - Hospital Foch, Suresnes
  - Institut Claudius Regaud, Toulouse
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Germany (15):
  - Urologicum Duisburg, Duisburg
  - Centrum fur Hamatologie und Onkologie Bethanien, Frankfurt
  - Universitätsklinikum Frankfurt, Klinik für Urologie, Frankfurt
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - Marien Hospital Herne, Herne
  - Universitatsklinikum Jena, Jena
  - Institut für Versorgungsforschung in der Onkologie, Koblenz
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Mainz
  - Klinikum rechts der Isar der Technischen Universität München, Urologische Klinik und Poloklinik, München
  - Universitatsklinikum Munster, Klinik fur Urologie und Kinderurologie, Münster
  - Universitat Regensburg, Regensburg
  - Universitatsklinikum Tubingen, Klinik fur Urologie, Tübingen
- Greece (5):
  - Henry Dunant Hospital Center, 4th Oncology Department, Athens
  - University General Hospital of Ioannina, Oncology Department, Ioannina
  - Athens Medical Center, Oncology Department, Marousi
  - General Hospital of Patras Agios Andreas, Pátrai
  - Anassa General Clinic, Oncology-Chemotherapy Department, Volos
- Italy (13):
  - Ospedale San Donato, Arezzo
  - Centro di Riferimento Oncologico IRCCS, Aviano
  - ASST Cremona, Cremona
  - Ospedale Policlinico San Martino IRCCS, Genoa
  - Istituto Romagnolo per Io Studio dei Tumori (IRST) "Dino Amadori", Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Maggiore della Carita, Novara
  - Istituto Oncologico Veneto IRCCS - Ospedale Busonera, Padua
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Instituto Nazionale Tumori Regina Elena - IFO, Roma
  - Azienda Ospedaliera Santa Maria di Temi, Terni
  - Centro Ricerche Cliniche di Verona srl, Verona
- South Korea (14):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Chonnam National University Hospital, Gwangju
  - Chonnam National University Hwasun Hospital, Hwasun
  - Korea University - Anam Hospital, Seongbuk-Gu
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - Yonsei University - Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (18):
  - Institut Catala d'Oncologia Badalona - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - CEIC Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas
  - MD Anderson Cancer Centre, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puera de Hierro Majadahonda, Majadahonda
  - Hospital Sant Joan de Deu, Manresa
  - Complejo Hospitalario de Ourense, Ourense
  - Hospital Universitario Marques de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Turkey (Türkiye) (8):
  - Ankara Sehir Hastanesi, Ankara
  - Dicle Universitesi Tip Fakultesi Hastanesi, Diyarbakır
  - Trakya Universitesi Saglik Arastirma ve Uygulama Merkezi, Edrine
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi Hastanesi, Istanbul
  - Medipol Mega Universite Hastanesi, Istanbul
  - T.C. Saglik Bakanligi Goztepe Prof Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Izmir Medical Point Hastanesi, Medikal Onkoloji Departmant, Izmir
  - Baskent Universitesi Adana Dr.Turgut Noyan Uygulama ve Arastima Merkezi, Seyhan
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Barts Health NHS Trust, London
  - East and North Hertfordshire NHS Trust, Northwood
  - The Royal Marsden NHS Foundation Trust, Surrey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petrylak DP, Tagawa ST, Jain RK, Bupathi M, Balar A, Kalebasty AR, George S, Palmbos P, Nordquist L, Davis N, Ramamurthy C, Sternberg CN, Loriot Y, Agarwal N, Park C, Tonelli J, Vance M, Zhou H, Grivas P. TROPHY-U-01 Cohort 2: A Phase II Study of Sacituzumab Govitecan in Cisplatin-Ineligible Patients With Metastatic Urothelial Cancer Progressing After Previous Checkpoint Inhibitor Therapy. J Clin Oncol. 2024 Oct 10;42(29):3410-3420. doi: 10.1200/JCO.23.01720. Epub 2024 Aug 26. PMID 39186707
- [Derived] Loriot Y, Kalebasty AR, Flechon A, Jain RK, Gupta S, Bupathi M, Beuzeboc P, Palmbos P, Balar AV, Kyriakopoulos CE, Pouessel D, Sternberg CN, Tonelli J, Sierecki M, Zhou H, Grivas P, Barthelemy P, Bangs R, Tagawa ST. A plain language summary of the TROPHY-U-01 study: sacituzumab govitecan use in people with locally advanced or metastatic urothelial cancer. Future Oncol. 2024;20(23):1621-1631. doi: 10.2217/fon-2023-1030. Epub 2024 Jun 5. PMID 38682560
- [Derived] Grivas P, Pouessel D, Park CH, Barthelemy P, Bupathi M, Petrylak DP, Agarwal N, Gupta S, Flechon A, Ramamurthy C, Davis NB, Recio-Boiles A, Sternberg CN, Bhatia A, Pichardo C, Sierecki M, Tonelli J, Zhou H, Tagawa ST, Loriot Y. Sacituzumab Govitecan in Combination With Pembrolizumab for Patients With Metastatic Urothelial Cancer That Progressed After Platinum-Based Chemotherapy: TROPHY-U-01 Cohort 3. J Clin Oncol. 2024 Apr 20;42(12):1415-1425. doi: 10.1200/JCO.22.02835. Epub 2024 Jan 23. PMID 38261969
- [Derived] Tagawa ST, Balar AV, Petrylak DP, Kalebasty AR, Loriot Y, Flechon A, Jain RK, Agarwal N, Bupathi M, Barthelemy P, Beuzeboc P, Palmbos P, Kyriakopoulos CE, Pouessel D, Sternberg CN, Hong Q, Goswami T, Itri LM, Grivas P. TROPHY-U-01: A Phase II Open-Label Study of Sacituzumab Govitecan in Patients With Metastatic Urothelial Carcinoma Progressing After Platinum-Based Chemotherapy and Checkpoint Inhibitors. J Clin Oncol. 2021 Aug 1;39(22):2474-2485. doi: 10.1200/JCO.20.03489. Epub 2021 Apr 30. PMID 33929895
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT03547973